CLINICAL TRIAL: NCT01866956
Title: Computerized Screening for Comorbidity in Adolescents With Substance or Psychiatric Disorders
Status: Completed | Type: Observational
Sponsor: Center for Psychological Consultation (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Pittsburgh (Other); Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other); Child Mind Institute (Other)
Responsible Party: Principal Investigator, Kenneth A. Kobak, Ph.D., Owner, Center for Psychological Consultation
Other Study IDs: 1R43MH094092 (NIH); 1R43MH094092 (NIH)
Record Dates: First submitted 2013-05-29; First posted 2013-06-03 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Psychiatric Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The KSADS-COMP will facilitate identification of comorbid psychiatric and substance use diagnoses frequently missed in clinical practice, and improve adolescent treatment outcomes. The self-administered version of the KSADS-COMP can also be used cost-effectively in schools and juvenile justice settings where there is a growing interest in early identification and referral of youth in need of mental health services. The KSADS-Bridge assessment tool with its RDoC neurocognitive tasks, when completed with the self- or clinician administered KSADS-COMP, will help to create cross-talk between the DSM and RDoC diagnostic perspectives, and begin to generate a database on the relationship between RDoC constructs and treatment outcomes across a range of diagnostic categories.

DETAILED DESCRIPTION:
This Phase II SBIR grant is a follow-up to the Phase I SBIR grant "Computerized Screening for Comorbidity in Adolescents with Substance or Psychiatric Disorders." During Phase I, parent and adolescent self administered computerized versions of the psychiatric interview, the Kiddie Schedule for Affective Disorders and Schizophrenia (KSADS), were developed to assess DSM-IVR diagnoses in adolescents. Since the funding of the Phase I grant, there have been two significant developments in the field: the American Psychiatric Association's release of the DSM-5 manual, and NIMH's launch of the Research Domain Criteria (RDoC) initiative that aims to create the necessary database to derive a new psychiatric nomenclature informed by neuroscience, genetics, and psychology. The primary goals of Phase II include: 1) Update the parent and adolescent self-administered computerized KSADS (KSADS-COMP) so it is compatible with DSM-5 criteria; 2) Develop software for a clinician-administered computerized KSADS (KSADS-COMP); 3) Create a KSADS- Bridge product that includes a battery of RDoC computerized neurocognitive tasks that can be completed with the self- or clinician-administered KSADS-COMP; and 4) Examine the criterion, convergent, and discriminant validity of the self-administered KSADS-COMP, and the relationship among DSM-5 diagnoses, dimensional measures of psychopathology, and performance on RDoC neurocognitive tasks. Ultimately the aim of this initiative is to create an instrument that, in addition to providing a reliable comprehensive assessment tool for psychiatric disorders in adolescents, can bridge DSM-5 and RDoC diagnostic perspectives. A sample of 400 adolescents and their parents will be recruited for this study: half will complete the self-administered KSADS-COMP; the other half will complete the clinician-administered KSADSCOMP. All 400 adolescents and their parents, in addition to completing one of the KSADS-COMP versions, will also complete a battery of dimensional symptom rating scales. A subset of 210 adolescents and their parents will then complete the other version of the KSADS-COMP to test diagnostic concordance between the self- and clinician-administered KSADS-COMP. To obtain reliable Kappa estimates, this subset will include 30 adolescents with no psychopathology and 30 adolescents that meet criteria for each of the following diagnoses: conduct disorder, major depression, bipolar; substance use disorders; post traumatic stress disorder; and attention deficit hyperactivity disorder. This subset of 210 adolescents will also be administered the RDoC battery of neurocognitive computerized tasks. The KSADS-COMP and KSADS-Bridge assessment tools will have multiple clinical and research applications. In addition to helping identify comorbidity in teens with substance or psychiatric disorders, it will help to create the cross-talk needed between the DSM and RDoC diagnostic perspectives, and will help to improve clinical care in the short- and long-run as the field aims to transition to a new psychiatric nomenclature.

ELIGIBILITY:
Inclusion Criteria:

* adolescent between the ages of 11 and 17

Exclusion Criteria:

* Children will be excluded if they have a diagnosis of mental retardation (IQ < 70) or a severe psychosis that would impair the child's ability to participate.

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: adolescents aged 13-18 seeking psychiatric treatment at a rural mental health clinic
Sampling Method: Non-Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Wilcoxon rank sum tests. | within 2 days of criterion measure
  compare scores on disorder-specific symptom rating scales between those with and without a specific diagnoses

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Hugo W. Moser Research Institute at Kennedy Krieger, Baltimore, Maryland
  - University of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Townsend L, Kobak K, Kearney C, Milham M, Andreotti C, Escalera J, Alexander L, Gill MK, Birmaher B, Sylvester R, Rice D, Deep A, Kaufman J. Development of Three Web-Based Computerized Versions of the Kiddie Schedule for Affective Disorders and Schizophrenia Child Psychiatric Diagnostic Interview: Preliminary Validity Data. J Am Acad Child Adolesc Psychiatry. 2020 Feb;59(2):309-325. doi: 10.1016/j.jaac.2019.05.009. Epub 2019 May 18. PMID 31108163